CLINICAL TRIAL: NCT05350241
Title: Exploring Temporospatial Gait Asymmetry, Dynamic Balance, and Locomotor Capacity After a 12-month Split-belt Treadmill Training in Adolescents With Unilateral Cerebral Palsy: A Randomized Clinical Study
Brief Title: Repetitive Split-Belt Treadmill Perturbation in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0017
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-belt treadmill walking group (Experimental): Participants in this group performed repeated split-belt treadmill training with an error-augmentation strategy.
  Interventions: Other: Split-belt treadmill training
- Control group (Active Comparator): Participants in this group received the standard physical rehabilitation program
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Split-belt treadmill training — Participants in the split-belt walking group (experimental group) performed repeated split-belt treadmill training with an error-augmentation strategy (exaggeration of the initial step-length asymmetry) for 60 minutes, three times per week for 12 successive weeks. The training was conducted under close supervision of a licensed pediatric physical therapist according to safety performance guidelines defined by the American Academy of Pediatrics.
  Arms: Split-belt treadmill walking group
Other: Standard physical therapy — Participants in the control group received the standard physical therapy program. Each session lasted for 60 minutes, repeated three times a week, over 12 consecutive weeks. The program consisted of advanced balance training, gait training, postural and flexibility exercises, and strength training exercises.
  Arms: Control group

SUMMARY:
This study was designed to investigate the effect of repeated split-belt treadmill waking practice on gait symmetry, dynamic balance control, and locomotor capacity in adolescents with unilateral cerebral palsy (ULCP). Fifty-two children with ULCP were randomly allocated to the split-belt treadmill walking (n = 26; undergone split-elt treadmill training or the Control group (n =23, received standard rehabilitation program). Both groups were assessed for gait symmetry, dynamic balance control, and locomotor capacity pre and post-treatment.

DETAILED DESCRIPTION:
Fifty-two children with ULCP were recruited from the Physical Therapy Outpatient Clinic of the College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 10 and 16 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity levels 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, had attentional neglect, and if they had cardiopulmonary problems that could be exacerbated by exercise.

Outcome measures

1. Gait-symmetry Indices: Gait symmetry indices (Spatial and temporal) were measured through the portable GAITRite system.
2. Dynamic balance: The directional dynamic limit of stability (forward, backward, paretic, and non-paretic) and overall limit of stability were assessed using the Biodex balance system.
3. Locomotor capacity: This was assessed through the 6-minute walk test (6-MWT), the Timed Up and Down Stair test (TUDS), and the 10-meter Shuttle Run Test (10mSRT).

Both groups were trained for one hour, three times a week, for 12 successive weeks. The split-belt treadmill walking group performed repetitive split-belt treadmill training with an error-augmentation strategy (i.e., exaggeration of the initial step-length asymmetry). The control group received the standard rehabilitation program, which comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* Age 10-16 years
* Motor function level I or II according to the Gross Motor Function Classification System.
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities/contractures
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders that could be exacerbated by exercise.
* Perceptual and/or behavioral disorders.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Spatial gait asymmetry index | 2 months
  The spatial gait asymmetry index was measured about the step length of the paretic and non-paretic leg through the portable GAITRite system. Lower scores indicate a more symmetrical pattern.
Temporal gait asymmetry index | 2 months
  was measured about the single-limb support time of the paretic and non-paretic leg The temporal gait asymmetry index through the portable GAITRite system. Lower scores indicate a more symmetrical pattern.
Dynamic limit of postural stability | 2 months
  The capacity to control and move the center of gravity in various directions across their base of support was assessed utilizing the Biodex balance system. Values are expressed as accuracy % and higher scores mean better balance capability.

SECONDARY OUTCOMES:
Six-minute walk test | 2 months
  The six-minute walk test measured the walking distance that children were able to cover across a 30-m walkway with a self-determined walking pace over six minutes. A longer distance indicates a better performance.
Timed Up and Down Stair test | 2 months
  The Timed Up and Down Stair test assessed the capacity (as time in seconds) to walk up and down a stair flight (14 steps, each was 20-cm in height). A shorter time to complete indicates better performance.
10-meter Shuttle Run Test | 2 months
  The 10-meter Shuttle Run Test measured the children's ability to walk and run at a faster rate. The test was performed twice over a 10-m path, and the better (faster) trial was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No